CLINICAL TRIAL: NCT05787652
Title: An Online Self-regulation Intervention to Support Weight Loss Among Adults Living With Obesity: a Randomised Controlled Trial
Brief Title: Adults Regulating Their Weight Everyday With Mobile Internet Support
Acronym: ARTEMIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute of Health and Care Research, United Kingdom (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARTEMIS
Record Dates: First submitted 2023-02-28; First posted 2023-03-28 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Obesity
Keywords: Obesity; Digital intervention; Mobile app; Self-regulation; Weight loss
MeSH Terms: conditions — Obesity; Self-Control; Weight Loss

STUDY DESIGN:
Intervention Model Description: This is a parallel group, randomised, controlled superiority trial.
Masking Description: It will not be possible to blind participants or trial staff to treatment allocation, as the control group receives no intervention and participants will be aware of the general nature of the study. However, all follow-up is done remotely and will therefore be unbiased.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARTEMIS mobile app (Experimental): Intervention participants will be asked to download the ARTEMIS app in the Apple or Google Play app stores. The app will comprise of daily self-weighing, daily weight-recording, daily action-planning, and weekly reports and reflection. Daily weight loss action plans will predominantly relate to diet, physical activity and sleep, and comprise of eight categories, to be chosen by participants and rotated on a weekly basis, each with 5-10 actions, to be chosen by participants and rotated on a daily basis. Participants can explore and engage in all of these actions for as long as they wish within the 26-weeks of the intervention but will be recommended to continue within the 'active exploratory phase' of the intervention for at least four weeks, before moving to a 'maintenance phase', where participants continue with the actions which worked best for them in the 'active exploratory phase'.
  Interventions: Behavioral: ARTEMIS mobile app
- Control (No Intervention): Control group participants will receive no intervention. They will be thanked for taking part in the study, advised that they may want to lose weight on their own and reminded of the next assessment at 12 weeks. The investigators will explain the value of control groups in randomised trials and the impact that remaining in follow-up has for the impact of the trial. They will also be reminded that they will receive equal financial reimbursement.

INTERVENTIONS:
Behavioral: ARTEMIS mobile app — Access to a self-regulation based mobile application.
  Arms: ARTEMIS mobile app

SUMMARY:
Adults Regulating Their weight Everyday with Mobile Internet Support (ARTEMIS) is a randomised controlled trial evaluating the effectiveness of a mobile app based weight loss intervention designed to increase self-regulation in adults living with obesity.

DETAILED DESCRIPTION:
Adults Regulating Their weight Everyday with Mobile Internet Support (ARTEMIS) is a randomised, controlled trial examining the effectiveness of the self-regulation intervention to promote weight loss, when delivered through a mobile application, with no in-person contact, among a sample of ~ 1,294 adults living with obesity in the United Kingdom. Further, the investigators will assess the safety of the intervention regarding any a potential unintended consequence, which is the development of disordered eating. The intervention comprises daily self-weighing and daily reflection on the day's task of controlling weight through implementation of actions, and selection of new actions for the next day. It encourages users to build up a repertoire of actions for life that suit them in controlling weight.

ELIGIBILITY:
Participation is open to those who meet the following eligibility criteria:

* aged ≥ 18 years;
* living with obesity (BMI ≥ 30 if of white ethnicity; ≥ 27.5 for all other ethnic groups);
* full- time residents in the UK, without the intention to move outside the UK within the next 12 months;
* able to access the internet with a smartphone;
* able to access and use a digital weighing scale;
* can understand English;
* not presently signed up with an intention to attend, or have in the previous three months attended, a weight management programme;
* not currently participating in another weight management study;
* not lost > 5 kg (10 pounds) body weight in the previous six months;
* not undergone bariatric surgery, or presently scheduled to have bariatric surgery;
* not pregnant, or planning a pregnancy in the next 12 months;
* not previously been diagnosed with an eating disorder;
* not recently been diagnosed with a disease, or expected to undergo treatment for a disease, associated with substantial weight loss e.g., cancer treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1294 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2025-03-23 (Estimated); Study Completion 2025-03-23 (Estimated)

PRIMARY OUTCOMES:
Change in body weight | 6 months (baseline to 26-week follow up)
  To assess if the intervention achieves significantly greater weight loss than the no-treatment control group.
Proportion of participants achieving ≥ 5% loss in body weight | 6 months (baseline to 26-week follow up)
  To assess if the intervention achieves significantly greater weight loss than the no-treatment control group.

SECONDARY OUTCOMES:
Change in body weight | 12 weeks (baseline to 12-week follow up)
  To assess if the intervention achieves significantly greater weight loss than the no-treatment control group in the short term.
Proportion of participants achieving ≥ 5% loss in body weight | 12 weeks (baseline to 12-week follow up)
  To assess if the intervention achieves significantly greater weight loss than the no-treatment control group in the short term.
Change in the proportion of participants scoring above threshold (> 7) on a modified Eating Disorders Examination - Questionnaire Short Form (EDE-QS) | 12- and 26-week follow up (baseline to 12 and 26-week follow up)
  To assess the impact of self-regulation intervention on disordered weight control. Note. the modified Eating Disorders Examination - Questionnaire Short Form (EDE-QS) has a maximum score of 18, with higher scores being indicative of disordered eating.

OTHER OUTCOMES:
Number of days with any app engagement | 26 weeks
  Process measure to assess whether the intervention engaged participants.
Number of daily weight readings | 26 weeks
  This is a process measure to assess whether the intervention engaged participants. This will be assessed as: 1. the total number of action plans completed; 2) the total number of action plans completed vs the total number of action plans selected, within the ARTEMIS app.
Number of daily actions selected | 26 weeks
  This is a process measure to assess whether the intervention engaged participants. This will be assessed as: 1. the total number of action plans completed; 2) the total number of action plans completed vs the total number of action plans selected, within the ARTEMIS app.
Number of daily action plans | 26 weeks
  This is a process measure to assess whether the intervention engaged participants. This will be assessed as: 1. the total number of action plans completed; 2) the total number of action plans completed vs the total number of action plans selected, within the ARTEMIS app.
Number of weekly reflections completed | 26 weeks
  This is a process measure to assess whether the intervention engaged participants. This will be assessed as: 1. the total number of action plans completed; 2) the total number of action plans completed vs the total number of action plans selected, within the ARTEMIS app.
Percentage of actions successfully completed | 26 weeks
  This is a process measure to assess whether the intervention engaged participants. This will be assessed as: 1. the total number of action plans completed; 2) the total number of action plans completed vs the total number of action plans selected, within the ARTEMIS app.
Self report of other weight management programmes accessed (purpose built questionnaire) | 12 and 26 weeks
  This is a process measure to assess whether the intervention led to participants taking action to manage their weight. This will be assessed using a purpose build questionnaire which asks participants "1.Have you taken any actions to manage your weight since the last assessment?". If Yes to question 1, this questionnaire further asks the following "2. What have you being doing to manage your weight (please click all that apply): Actively using the ARTEMIS app; using learned strategies from the ARTEMIS app, but not actively using app; using another online or app based weight loss programme; attending a weight loss programme where I see someone face-to-face; using weight loss medication; using a meal replacement programme; other (please specify further in the text box below).
Perceived barriers contributing to non-completion of daily action plans | 26 weeks
  This is a process measure to assess whether the intervention engaged participants. This will be recorded by participants entering free text into the app once prompted when they have indicated they have not completed their daily action plan i.e., "Please tell us why were you unable to perform your action yesterday? Is there anything you think would be useful to do differently next time you choose this action?". The investigators will use content analysis to analyse these data.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Aveyard, PhD, Principal Investigator — University of Oxford
Locations (1):
- Online social media platforms (Meta (Facebook, Instagram, Google, Twitter), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doody P, Wren GM, Mounsey S, Haasova S, Stewart C, Haffner SJP, Jebb SA, Aveyard P. The effectiveness and safety of a mobile application-based self-regulation intervention to support weight loss among adults living with obesity: a large-scale pragmatic randomised controlled trial. BMC Med. 2025 Nov 29;24(1):6. doi: 10.1186/s12916-025-04519-8. PMID 41316243

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-06-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT05787652/SAP_001.pdf